CLINICAL TRIAL: NCT01072773
Title: Phase II Study of Bortezomib, Cyclophosphamide and Dexamethasone in Patients With Primary Systemic Light Chain Amyloidosis
Brief Title: Bortezomib, Cyclophosphamide, and Dexamethasone in Treating Patients With Primary Systemic Light Chain Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0985; NCI-2009-01564 (Registry Identifier: NCI's CTRP); 09-005736 (Other: Mayo Clinic IRB); MC0985 (Other: Mayo Clinic Cancer Center); X05306 (Other: MPI Protocol)
Record Dates: First submitted 2010-02-17; First posted 2010-02-22 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Primary Systemic Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Bortezomib; Cyclophosphamide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortez/Cyc/Dex (Experimental): Bortezomib IV on days 1, 8, and 15, oral cyclophosphamide and oral dexamethasone once daily on days 1, 8, 15, and 22.
  Interventions: Drug: bortezomib; Drug: cyclophosphamide; Drug: dexamethasone

INTERVENTIONS:
Drug: bortezomib — 1.3 mg/m^2, by IV on days 1, 8 and 15 every 28 days
  Other Names: LDP 341; MLN341; PS-341; VELCADE
Drug: cyclophosphamide — 300 mg/m^2, orally, on days 1, 8, 15 & 22 every 28 days.
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Drug: dexamethasone — 40 mg, orally, on days 1, 8, 15 & 22 every 28 days
  Other Names: Aeroseb-Dex; Decaderm; Decadron; Decaspray; DM; DXM

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib, cyclophosphamide, and dexamethasone together works in treating patients with primary systemic light chain amyloidosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the confirmed hematologic response rate of the combination of bortezomib, cyclophosphamide and dexamethasone in patients with primary systemic amyloidosis.

SECONDARY OBJECTIVES:

I. Organ response rate of the bortezomib, cyclophosphamide and dexamethasone combination.

II. Severity and frequency of adverse events associated with bortezomib, cyclophosphamide and dexamethasone treatment in patients with primary systemic amyloidosis.

III. Time to progression.

IV. Survival.

OUTLINE: Patients receive bortezomib IV on days 1, 8, and 15 and oral cyclophosphamide and oral dexamethasone once daily on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histochemical diagnosis of amyloidosis as based on detection by polarizing microscopy of green birefringent material in Congo red-stained tissue specimens
* Measurable disease of amyloid light chain amyloidosis as defined by at least ONE of the following: serum monoclonal protein >= 1.0 g by protein electrophoresis, > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis, serum free light-chain >= 7.5 mg/dL with an abnormal kappa:lambda ratio
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2
* Absolute neutrophil count >= 1000/uL
* Platelet >= 75000/uL
* Total bilirubin < 3.0 mg/dL
* Aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Creatinine clearance >= 30ml/min
* Women of childbearing potential should have a negative serum or urine pregnancy test done =< 7 days prior to registration, and should be willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Male subject agrees to use an acceptable method for contraception for the duration of the study
* Previously treated amyloidosis; no limit to prior therapy provided there is adequate residual organ function
* Symptomatic organ involvement (heart, kidney, liver/GI tract, peripheral nervous system or soft tissue); carpal tunnel syndrome skin purpura, or the presence of vascular amyloid on a bone marrow biopsy alone are not sufficient to meet criteria for "symptomatic organ involvement"
* Renal involvement is defined as proteinuria (predominantly albumin) > 0.5 g/day in a 24- hour urine collection
* Cardiac involvement is defined as the presence of a mean left ventricular wall thickness on echocardiogram greater than 12 mm in the absence of a history of hypertension or valvular heart disease, or in the presence of unexplained low voltage (< 0.5 mV) on the electrocardiogram
* Hepatic involvement is defined as hepatomegaly (>= 2 cm below costal margin) on physical exam or an alkaline phosphatase > 1.5 x ULN
* Peripheral nerve involvement is defined based on clinical history or abnormal sensory and/or motor findings on neurologic exam
* Autonomic nerve involvement is defined as orthostasis, symptoms of nausea or dysgeusia, gastric atony by gastric emptying scan, diarrhea or constipation
* Soft tissue and lymphatic involvement may be ascertained based on classic physical exam findings (macroglossia, shoulder pad sign, raccoon eyes, carpal tunnel syndrome, synovial enlargement, firm enlarged lymph nodes) or biopsy
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by subject any time without prejudice to future medical care
* Willingness to return to Mayo Clinic enrolling institution for follow-up

Exclusion Criteria:

* Melphalan or other myelosuppressive agents =< 3 weeks prior to registration; non-myelosuppressive agents like thalidomide, or high dose corticosteroids <= 1week prior to registration
* Concurrent use of corticosteroids, but patients may be on chronic steroids (maximum dose 20 mg/day prednisone equivalent) if they are being given for disorders other than amyloid, i.e., adrenal insufficiency, rheumatoid arthritis, etc
* Any of the following because this study involves an agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown: pregnant women and nursing women
* Other active malignancy =< 2 years prior to registration; EXCEPTIONS: Nonmelanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: If there is a history or prior malignancy, they must not be receiving any specific treatment for their cancer
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens including psychiatric illness/social situations that would limit compliance with study requirements
* Known to be HIV positive
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Clinically overt multiple myeloma (monoclonal Bone Marrow Plasma Count > 30%), and at least one of the following: bone lesions or hypercalcemia
* History of myocardial infarction =< 6 months, or requiring use of ongoing maintenance drug therapy for life-threatening ventricular arrhythmias
* Grade 3 sensory or grade 1 painful peripheral neuropathy
* Known hypersensitivity to bortezomib, boron or mannitol
* Cardiac syncope, uncompensated New York Heart Association (NYHA) Class 3 or 4 congestive heart failure or troponin T > 0.1 ng/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bortez/Cyc/Dex
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bortez/Cyc/Dex
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 69 [67 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
Prior Treatment [Mean (Full Range); unit: Prior Treatments] — Number of previous regimens used for the treatment of amyloidosis. There is no limit to the number of prior therapies provided there is adequate residual organ function.
  Prior Treatments | 6.5 [1 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Confirmed Hematologic Response
Description: Response that was confirmed on 2 consecutive evaluations during treatment.
  Complete Response(CR): Complete disappearance of M-protein from serum and urine on immunofixation, normalization of Free Light Chain (FLC) ratio and <5% plasma cells in bone marrow.
  Very Good Partial Response(VGPR): >=90% reduction in serum M-component; Urine M-Component <=100 mg per 24 hours.
  Partial Response(PR): >=50% reduction in serum M-component and/or Urine M-Component >=90% reduction or <200 mg per 24 hours; or >=50% decrease in difference between involved and uninvolved FLC levels.
Time Frame: Duration of treatment (up to 12 cycles/months)
Measure: Number; unit: participants
Arm/Group | Bortez/Cyc/Dex
Number analyzed (Participants) | 2
participants
  Complete Response (CR) | 0
  Very Good Partial Response (VGPR) | 0
  Partial Response (PR) | 0

2. Secondary Outcome: Number of Participants With Treatment Related Adverse Events.
Description: Adverse events (AE) that are classified as either possibly, probably, or definitely related to study treatment according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE version 3.0). The maximum grade for each type of AE will be recorded for each patient. Grade refers to the severity of the AE.
  Grade 1: Mild AE, Grade 2: Moderate AE, Grade 3: Severe AE, Grade 4: Life-threatening or disabling AE, Grade 5: Death related AE
  Adverse events will be assessed using NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0.
Time Frame: Duration on treatment (up to 12 cycles/months)
Measure: Number; unit: participants
Arm/Group | Bortez/Cyc/Dex
Number analyzed (Participants) | 2
participants
  Grade 1-2 | 2
  Grade 3-4 | 0
  Grade 5 | 0

3. Secondary Outcome: Number of Participants With an Organ Response.
Description: The number of patients that acheived a response in an affected organ.
Time Frame: Duration on treatment (up to 12 cycles/months)
Measure: Number; unit: participants
Arm/Group | Bortez/Cyc/Dex
Number analyzed (Participants) | 2
participants | 0

4. Secondary Outcome: Overall Survival
Description: Survival time is defined as the time from registration to death due to any cause.
Time Frame: Duration of Study (up to 5 years)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bortez/Cyc/Dex
Number analyzed (Participants) | 2
Months | 1.45 [1.35 to 1.54]

5. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to the earliest date of documented disease progression. If a patient dies without a documentation of disease progression the patient will be considered to have had tumor progression at the time of their death
Time Frame: Duration of Study (up to 5 years)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bortez/Cyc/Dex
Number analyzed (Participants) | 2
Months | 1.45 [1.35 to 1.54]

6. Secondary Outcome: Duration of Response
Description: Duration of response will be calculated from the date of first evidence of response until the date of progression in the subset of patients with confirmed hematologic responses.
Time Frame: Duration of Study (up to 5 years)
Population: Neither participant achieved a response. Therefore, no duration of response calculation was performed.
Arm/Group | Bortez/Cyc/Dex
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Bortez/Cyc/Dex
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortez/Cyc/Dex (N=2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortez/Cyc/Dex (N=2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes